CLINICAL TRIAL: NCT01179295
Title: Phase 1 Study of Single Agent BAY86-9766 in Japanese Patients With Advanced or Refractory Solid Tumors
Brief Title: Japanese BAY86-9766 Monotherapy Phase I Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15091
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Neoplasms
Keywords: MEK inhibitor; BAY86-9766; RDEA 119; Solid tumor
MeSH Terms: conditions — Neoplasms | interventions — N-(3,4-difluoro-2-(2-fluoro-4-iodophenylamino)-6-methoxyphenyl)-1-(2,3-dihydroxypropyl)cyclopropane-1-sulfonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: BAY86-9766
- Arm 2 (Experimental)
  Interventions: Drug: BAY86-9766
- Arm 3 (Experimental)
  Interventions: Drug: BAY86-9766
- Arm 4 (Experimental)
  Interventions: Drug: BAY86-9766

INTERVENTIONS:
Drug: BAY86-9766 — BAY86-9766 30 mg twice a day (bid).
  Arms: Arm 1
Drug: BAY86-9766 — BAY86-9766 50 mg twice a day (bid).
  Arms: Arm 2
Drug: BAY86-9766 — BAY86-9766 100 mg once a day (od)
  Arms: Arm 3
Drug: BAY86-9766 — BAY86-9766 60 mg once a day (od)
  Arms: Arm 4

SUMMARY:
This is an uncontrolled, open-label, non-randomized phase I / pharmacokinetic study of oral BAY86-9766 to investigate the safety, tolerability, pharmacokinetics, and efficacy profiles in Japanese patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients, who are at least 18 years of age at the first screening examination/ visit, with advanced or refractory solid tumors not amenable to standard therapy.
* Histological or cytological documentation of non-hematologic, malignant solid tumor, excluding primary brain or spinal tumors, with no current involvement in the central nervous system (CNS)
* At least one measurable lesion or evaluable disease according to response evaluation criteria in solid tumors (RECIST) version 1.1
* Eastern cooperative oncology group performance status (ECOG-PS) of 0 or 1
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Use of any anti-cancer therapy including chemotherapy, investigational agents or devices and immunotherapy within 4 weeks of the first dose of study medication
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management
* Known human immunodeficiency virus (HIV) infection or chronic active hepatitis B or C
* Inadequate bone marrow, liver and renal function
* Inability to swallow oral medications or any condition that could affect the absorption of orally administered drugs
* Concomitant treatment with cytochrome P450 isoenzymes CYP3A4 inhibitors/inducers, and CYP2C19 inhibitors/ inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11-19 (Actual); Primary Completion 2012-04-27 (Actual); Study Completion 2012-04-27 (Actual)

PRIMARY OUTCOMES:
Safety evaluation due to results of physical examinations, vital signs, AEs, abnormal laboratory tests and 12-lead ECG, cardiac function test and ophthalmological examination. | At the end of 30-day follow up after discontinuation of study drug administration
Calculation of pharmacokinetic parameters of BAY86-9766 and its metabolite (M17). | Cycle 1 Day 22 and Day 23 for Cohorts 1 & 2 and Cohorts 3 & 4, respectively.

SECONDARY OUTCOMES:
Response rate | On average 3 months
Disease control rate | On average 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Kashiwa, Chiba, Japan